CLINICAL TRIAL: NCT03396354
Title: Prospective Comparison of Surgical Outcomes With Using Integrated Robotic Technology Versus Conventional Laparoscopy for Gastric Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-1066
Record Dates: First submitted 2018-01-04; First posted 2018-01-10 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Gastric Cancer Patients Undergoing Minimally Invasive Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated robotic surgery (Experimental)
  Interventions: Procedure: Integrated robotic surgery
- Conventional laparoscopic surgery (Active Comparator)
  Interventions: Procedure: Conventional laparoscopic surgery

INTERVENTIONS:
Procedure: Integrated robotic surgery — Robotic gastrectomy using Single-Site and Firefly technology will be performed. Specifically, two-port surgery using the Single-Site port and an independent trocar along the right flank (for harmonic scalpel) will be used, along with peritumoral injection of indocyanine green via endoscopy the day before surgery to completely visualize the entire lymphatic channel.
  Arms: Integrated robotic surgery
Procedure: Conventional laparoscopic surgery — conventional laparoscopic gastrectomy will be performed.
  Arms: Conventional laparoscopic surgery

SUMMARY:
Despite the theoretical superiority of robotic technology, surgical outcomes following robotic surgery have shown little benefit over conventional laparoscopic surgery. At present, studies have evaluated the value of robotic technology in clinical practice, including EndoWrist®, TilePro®, Firefly®, and Single-Site®, and have demonstrated the possibility of added clinical value, specifically in regards to decreased postoperative pancreatic fistula, usefulness as a multi-display education system, visualization of lymphatic channels, and implementation of reduced-port robotic gastrectomy. However, these technologies have only been applied independently and not in a well-organized manner.

Maximizing radicality and safety while minimizing invasiveness are critical to bettering cancer surgery. We hypothesize that robot technology can affect these factors positively and that the use of appropriate parameters thereof could help shed more light on the benefits of a robotic system in gastric cancer surgery.

1. Radicality: added benefit of Firefly® for lymph node visualization Number of retrieved lymph nodes can be considered a surrogate marker of long-term survival. In our proposed study, we will focus on the number of retrieved (lymph nodes as the primary outcome. Additionally, bleeding, which is known to be associated with poor overall survival, will be measured as a secondary outcome. Three-year recurrence free survival and 5-year overall survival will be followed up.
2. Safety: benefit of Firefly® in differentiating lymph nodes from other organs and benefit of a magnified view and EndoWrist® Although robotic surgery reportedly shows less in-hospital and outpatient complication rates, a higher number of enrolled patients is needed to statistically validate these results. In the currently proposed study, these would be secondary outcomes. We have experienced the benefit of using fluorescence imaging to differentiate lymph node from biliary trees and pancreas parenchyma. As a reflection thereof, bleeding would be measured as parameter of unintended injury to a normal organ. To evaluate injury to pancreas parenchyma and postoperative pancreatic fistula, amylase/lipase levels in serum and drainage fluid will be measured.
3. Invasiveness: value of Single-Site® Serum CRP (C reactive protein) levels (day 0, day 3, day 5, and 4 weeks after surgery) and pain scores (at 6 hr, 12 hr, 24 hr, 48 hr, and 72 hr after surgery) will be measured to evaluate surgical trauma to the patients. Satisfaction on the wound will be evaluated using Korean version of the body image scale at one month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of gastric adenocarcinoma and scheduled to undergo minimally invasive gastrectomy
* Age > 20 years
* A patient who signed the informed consent

Exclusion Criteria:

* Mentally incompetent, illiterate, or pregnant patients
* Requiring major combined resection (colon, pancreas, etc., except the gall bladder)
* Having metastatic or non-resectable lesion.
* Active other cancer history

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
Number of retrieved LN | during the gastrectomy surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea

REFERENCES:
- [Background] Kim HI, Han SU, Yang HK, Kim YW, Lee HJ, Ryu KW, Park JM, An JY, Kim MC, Park S, Song KY, Oh SJ, Kong SH, Suh BJ, Yang DH, Ha TK, Kim YN, Hyung WJ. Multicenter Prospective Comparative Study of Robotic Versus Laparoscopic Gastrectomy for Gastric Adenocarcinoma. Ann Surg. 2016 Jan;263(1):103-9. doi: 10.1097/SLA.0000000000001249. PMID 26020107
- [Background] Zeng YK, Yang ZL, Peng JS, Lin HS, Cai L. Laparoscopy-assisted versus open distal gastrectomy for early gastric cancer: evidence from randomized and nonrandomized clinical trials. Ann Surg. 2012 Jul;256(1):39-52. doi: 10.1097/SLA.0b013e3182583e2e. PMID 22664559
- [Background] Vizza E, Corrado G, Mancini E, Baiocco E, Patrizi L, Fabrizi L, Colantonio L, Cimino M, Sindico S, Forastiere E. Robotic single-site hysterectomy in low risk endometrial cancer: a pilot study. Ann Surg Oncol. 2013 Aug;20(8):2759-64. doi: 10.1245/s10434-013-2922-9. Epub 2013 Mar 7. PMID 23468046
- [Background] Kim HH, Hyung WJ, Cho GS, Kim MC, Han SU, Kim W, Ryu SW, Lee HJ, Song KY. Morbidity and mortality of laparoscopic gastrectomy versus open gastrectomy for gastric cancer: an interim report--a phase III multicenter, prospective, randomized Trial (KLASS Trial). Ann Surg. 2010 Mar;251(3):417-20. doi: 10.1097/SLA.0b013e3181cc8f6b. PMID 20160637
- [Background] Pietrabissa A, Sbrana F, Morelli L, Badessi F, Pugliese L, Vinci A, Klersy C, Spinoglio G. Overcoming the challenges of single-incision cholecystectomy with robotic single-site technology. Arch Surg. 2012 Aug;147(8):709-14. doi: 10.1001/archsurg.2012.508. PMID 22508669
- [Background] Kim YM, Baek SE, Lim JS, Hyung WJ. Clinical application of image-enhanced minimally invasive robotic surgery for gastric cancer: a prospective observational study. J Gastrointest Surg. 2013 Feb;17(2):304-12. doi: 10.1007/s11605-012-2094-0. Epub 2012 Dec 1. PMID 23207683
- [Background] Lee S, Kim JK, Kim YN, Jang DS, Kim YM, Son T, Hyung WJ, Kim HI. Safety and feasibility of reduced-port robotic distal gastrectomy for gastric cancer: a phase I/II clinical trial. Surg Endosc. 2017 Oct;31(10):4002-4009. doi: 10.1007/s00464-017-5435-y. Epub 2017 Feb 15. PMID 28205030
- [Background] Kitano S, Iso Y, Moriyama M, Sugimachi K. Laparoscopy-assisted Billroth I gastrectomy. Surg Laparosc Endosc. 1994 Apr;4(2):146-8. PMID 8180768
- [Derived] Choi S, Kim NY, Kim YN, Park SH, Kim KY, Cho M, Kim YM, Hyung WJ, Kim HI. Fluorescence-guided Two-port Robotic Gastrectomy Versus Conventional Laparoscopic Gastrectomy: A Nonrandomized Controlled Trial. Ann Surg Open. 2023 Jul 26;4(3):e318. doi: 10.1097/AS9.0000000000000318. eCollection 2023 Sep. PMID 37746613